CLINICAL TRIAL: NCT04167111
Title: Pilot Study- Treat to Target Vitamin D in End Stage Renal Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid pandemic
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 0646-19-FB
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Subjects will be started on Vitamin D3 4000 per day or 2400 IU per day at baseline and based on 3 month 25(OH)D levels, will be adjusted to a different vitamin D dose if needed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D 4000 (Active Comparator): At baseline, if subjects 25(OH)D levels are 12-19.9, they will be started on 4000 IU per day.
  Interventions: Dietary Supplement: Cholecalciferol
- Vitamin D 2400 (Active Comparator): At baseline, if subjects 25(OH)D levels are 20-30, they will be started on 2400 IU per day.
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Vitamin D
  Other Names: Vitamin D3

SUMMARY:
Feasibility of dose adjustment to reach a 6 month 25-hydroxy vitamin D level of 35-50 ng/ml in end stage renal disease patients

DETAILED DESCRIPTION:
Pilot study to test the feasibility of adjusting doses based on a prespecified algorithm to reach a 6 month 25(OH)D level of 35-50 ng/ml in end stage renal disease patients.

ELIGIBILITY:
Inclusion Criteria:

* likely be able to complete the study, >3 months on hemodialysis, receiving standard of care through their nephrologist.

Exclusion Criteria:

* on peritoneal dialysis, allergy to vitamin D, liver disease, intestinal disorders that interfere with vitamin D absorption, taking vitamin D >800 IU per day, 25(OH)D level >30 ng/ml, glucocorticoids, anticonvulsants or drug therapies for osteoporosis, pregnancy.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
25(OH)D level | 6 months
  25(OH)D level

CONTACTS AND LOCATIONS:
Overall Officials: Laura Graeff-Armas, MD, MS, PhD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No